CLINICAL TRIAL: NCT02312011
Title: A Phase 1/2a Blinded, Placebo-Controlled Study to Assess the Safety, Tolerability, and Dose-range Finding of Multiple Ascending Doses of ISIS 598769 Administered Subcutaneously to Adult Patients With Myotonic Dystrophy Type 1
Brief Title: A Safety andTolerability Study of Multiple Doses of ISIS-DMPKRx in Adults With Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 598769-CS2
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Myotonic Dystrophy Type 1
Keywords: Myotonic Dystrophy; DM1; Adult onset; Neuromuscular Disease; DMPKRx
MeSH Terms: conditions — Myotonic Dystrophy; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IONIS-DMPKRx (Experimental): IONIS DMPKRx is administered subcutaneously over the course of 6 weeks for dose levels 1, 2, 3, 4, and 5.
  IONIS DMPKRx is administered subcutaneously over the course of 12 weeks for dose levels 4 or 5.
  Interventions: Drug: IONIS-DMPKRx
- Placebo (Placebo Comparator): A placebo is administered subcutaneously over the course of 6 weeks. A placebo is administered subcutaneously over the course of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS-DMPKRx — Drug
  Other Names: ISIS 598769
  Arms: IONIS-DMPKRx
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will test the safety, tolerability, and pharmacokinetics of multiple escalating doses of ISIS-DMPKRx administered subcutaneously to adult patients with DM1.

DETAILED DESCRIPTION:
This is a Phase 1/2a multicenter, blinded, placebo-controlled study of ISIS-DMPK Rx in adult patients with DM1.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements
2. Males or females aged 20 to 55 years old at the time of informed consent
3. Satisfy the following:

   1. Females: non-pregnant and non-lactating, surgically sterile, post menopausal, abstinent, or if engaged in sexual relations of child-bearing potential, subject is using an acceptable contraceptive method from the time of signing the informed consent until at least 14 weeks after the last dose of Study Drug.
   2. Males: surgically sterile, abstinent or if engaged in sexual relations with a female of child-bearing potential, the subject must be using an acceptable contraceptive method from the time of signing the informed consent form until at least 14 weeks after the last dose of Study Drug.
4. BMI <35.0 kg/m2
5. Genetic confirmation of DM1 with DMPK CTG repeat length ≥ 100
6. Onset of DM1 symptoms after the age of 12
7. Clinically apparent myotonia equivalent to hand opening time of at least 2 seconds, in the opinion of the Investigator
8. Ambulatory (orthoses allowed, canes and walkers not allowed) and able to walk at least 25 meters at screening

Exclusion Criteria:

1. Clinically significant abnormalities in medical history (e.g., previous acute coronary syndrome within 6 months of screening, major surgery within 3 months of screening) or physical examination
2. Clinically significant abnormalities in screening laboratory values that would render the subject unsuitable for inclusion
3. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
4. Unwilling or unable to comply with study procedures (e.g., muscle biopsies), including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator
5. Known history of or previous positive test for human immunodeficiency virus (HIV), hepatitis C, or chronic hepatitis B
6. Active malignancy or history within last 5 years, except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix that has been successfully treated, or pilomatricoma
7. Treatment with another investigational drug, biologic agent, or device within one month of screening, or 5 half-lives of investigational agent, whichever is longer; any history of previous treatment with an oligonucleotide (including siRNA)
8. Recent history of or current drug or alcohol abuse
9. History of bleeding tendency or ongoing oral anticoagulation
10. Developmental delay, intellectual disability, or significant behavioral neuropsychiatric manifestations
11. Thyroid dysfunction that is untreated (if on thyroid hormone replacement therapy, need to have adequate and stable replacement over the previous 6 months)
12. Implanted device for the treatment of cardiac problems (i.e., pacemaker or defibrillator)
13. Clinically significant abnormal ECG or echocardiogram, or significant symptoms of cardiac dysfunction at Screening
14. Have a seizure disorder
15. If being treated with testosterone, on a stable replacement dose (i.e., for hypogonadism)
16. Treatment with corticosteroids within 8 weeks prior to the first dose of Study Drug
17. History of hypersensitivity to local anesthetics to be used in the biopsy procedure or components thereof
18. Treatment with anti-myotonia medication within 30 days prior to screening. May include, but not be limited to: Phenytoin, Carbamazepine, Procainamide, Disopyramide, Nifedipine, Acetazolamide, Clomipramine, Imipramine, Amytriptiline, Taurine, Quinine, Mexiletine
19. Have any condition, which, in the opinion of the investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety (The number of participants with adverse events) | Participants will be followed for the duration of the study; an expected 24 - 32 weeks
  The number of participants with adverse events
Tolerability (The number of participants with adverse events) | Participants will be followed for the duration of the study; an expected 24 -32 weeks
  The number of participants with adverse events

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (Cmax, Tmax) | Plasma at 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hours after dosing.
  * the maximal observed plasma drug concentration (Cmax)
  * the time to reach Cmax (Tmax)
  * the area under the plasma concentration time curve from the time of the subcutaneous dose to the last collected sample (24 hours after dosing)
Urine Pharmacokinetics (Amount of drug excreted in the urine) | 0-24 hours post-dosing
  Amount of drug excreted in the urine

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Stanford University Medical Center, Stanford, California
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - The Ohio State University, Columbus, Ohio
  - Houston Methodist, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Thornton CA, Moxley RT 3rd, Eichinger K, Heatwole C, Mignon L, Arnold WD, Ashizawa T, Day JW, Dent G, Tanner MK, Duong T, Greene EP, Herbelin L, Johnson NE, King W, Kissel JT, Leung DG, Lott DJ, Norris DA, Pucillo EM, Schell W, Statland JM, Stinson N, Subramony SH, Xia S, Bishop KM, Bennett CF. Antisense oligonucleotide targeting DMPK in patients with myotonic dystrophy type 1: a multicentre, randomised, dose-escalation, placebo-controlled, phase 1/2a trial. Lancet Neurol. 2023 Mar;22(3):218-228. doi: 10.1016/S1474-4422(23)00001-7. PMID 36804094